CLINICAL TRIAL: NCT04958109
Title: Evaluation of Kisspeptin Glucose-Stimulated Insulin Secretion With Oral Glucose Tolerance Test
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, Harvard Reproductive Endocrine Sciences Center, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 267339; 5K23HD097296 (NIH); NCT02953834 (obsolete NCT alias)
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases | interventions — Glucose Tolerance Test; Kisspeptins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kisspeptin (Experimental): • Intravenous administration of kisspeptin 112-121 x 16 hours
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Drug: Kisspeptin
- Placebo (Placebo Comparator): • Intravenous administration of placebo x 16 hours
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Drug: Placebo

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — Administration of a 75 gm oral glucose tolerance test
Drug: Kisspeptin — Intravenous administration of kisspeptin 112-121 x 16 hours
  Arms: Kisspeptin
Drug: Placebo — Intravenous administration of Placebo 16 hours
  Arms: Placebo

SUMMARY:
The goal of this study is to understand how exogenous kisspeptin affects metabolism by evaluating responses to an oral glucose tolerance test

DETAILED DESCRIPTION:
Assignment: Each study subject will serve as their own control. The order of the visits will be randomized.

Delivery of Interventions:

* Prior to the study visit, subjects will undergo a review of their medical history and screening laboratories.
* During the inpatient study, the subjects will

  * Undergo a 16-hour kisspeptin infusion
  * Undergo an oral glucose tolerance test

ELIGIBILITY:
Inclusion Criteria:

History:

* over the age of 18,
* normal pubertal development
* stable weight for previous three months,
* normal body mass index (BMI between 18.5-25)
* regular menstrual cycles

Physical examination:

• systolic BP < 140 mm Hg, diastolic < 90 mm Hg

Laboratory studies: (per Massachusetts General Hospital reference ranges)

* normal hemoglobin
* hemoglobin A1C < 6.5%
* blood urea nitrogen, creatinine not elevated
* aspartate aminotransferase, alanine aminotransferase < 3x upper limit of normal

Exclusion Criteria:

* active illicit drug use,
* history of a medication reaction requiring emergency medical care,
* difficulty with blood draws.
* history of chronic disease, except well controlled thyroid disease,
* recent use of prescription medications which interfere with metabolism or reproduction (recent = within 5 half-lives of the drug). Use of levothyroxine or seasonal allergy medications is acceptable,
* history of diabetes in a first degree relative,
* use of contraceptive pills, patches or vaginal rings within last 4 weeks.
* hyperlipidemia by fasting lipid panel
* positive serum pregnancy test (for all women)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lippincott, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Boston area. 16 participants consented and were screened for eligibility between 10/2021 and 10/2022
Pre-assignment Details: There was no wash out or run in period. 4 individuals were found to be ineligible by criteria.
Groups:
- Kisspeptin, Then Placebo: Oral Glucose Tolerance Test (OGTT): Administration of a 75 gm oral glucose tolerance test
  Kisspeptin: Intravenous administration of kisspeptin 112-121 x 16 hours, with administration of OGTT at hour 12 After at least 2 weeks and up to 6 months, then Placebo: Intravenous administration of Placebo 16 hours, with administration of OGTT at hour 12
- Placebo, Then Kisspeptin: • Intravenous administration of placebo x 16 hours
  Oral Glucose Tolerance Test (OGTT): Administration of a 75 gm oral glucose tolerance test
  Placebo: Intravenous administration of Placebo 16 hours, with administration of OGTT at hour 12 After at least 2 weeks and up to 6 months, then Kisspeptin: Intravenous administration of kisspeptin 112-121 x 16 hours, with administration of OGTT at hour 12
Period: Overall Study
Arm/Group | Kisspeptin, Then Placebo | Placebo, Then Kisspeptin
Started | 4 | 7
Completed | 4 | 5
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kisspeptin | Placebo | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (6.8) | 26 (6.8) | 26 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: per Participant flow only 5 participants completed in each arm
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 4 | 7 | 11
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Oral Glucose Sensitivity Index (Kisspeptin-Placebo)
Description: Change in Oral glucose Sensitivity Index between kisspeptin and placebo arms in oral glucose tolerance test
Time Frame: 3 hours
Population: Individuals who completed both studies were evaluated
Measure: Mean (Standard Deviation); unit: ml min-1m-2
Arm/Group | Kisspeptin | Placebo
Number analyzed (Participants) | 9 | 9
ml min-1m-2 | 517 (70) | 521 (82)

ADVERSE EVENTS:
Time Frame: From time of study consent until study completion (approximately 5 months).
Description: All participants were asked about new health symptoms at each visit.
Groups:
- Kisspeptin: Oral Glucose Tolerance Test(OGTT): Administration of a 75 gm oral glucose tolerance test Kisspeptin: Intravenous administration of kisspeptin 112-121 x 16 hours, then at hour 12 OGTT
- Placebo: Oral Glucose Tolerance Test (OGTT): Administration of a 75 gm oral glucose tolerance test Placebo: Intravenous administration of Placebo 16 hours, then at hour 12 OGTT
Arm/Group | Kisspeptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 6/9 | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kisspeptin (N=9) | Placebo (N=9)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Subject reported typical breast pain associated with menstruation, while menstruating
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) — IV site reaction or bruise
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Subject reported menstrual cramps while menstruating
Irregular Menstruation (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Infections and Infestations - Other, Specify (Infections and infestations) | 1 (1) | 2 (2) — Coronavirus disease infection 2019 No subject had the Infection during active study protocol
Fatigue (General disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was designed as a pilot study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT04958109/Prot_SAP_000.pdf